CLINICAL TRIAL: NCT01029626
Title: Glasgow-Blatschford Score Validation for Stratification of Patients With Digestive Hemorrhage
Brief Title: Glasgow-Blatschford Score Validation in Digestive Hemorrhage
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Geneva (Other)
Responsible Party: Principal Investigator, Marc Girardin, MD, University Hospital, Geneva
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 09-091
Record Dates: First submitted 2009-12-09; First posted 2009-12-10 (Estimated); Last update posted 2018-06-01 (Actual); Status verified 2018-05

CONDITIONS: Gastrointestinal Hemorrhage
MeSH Terms: conditions — Gastrointestinal Hemorrhage | interventions — Endoscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Endoscopy (Other): If the Glasgow-Blatchford score is zero, the endoscopy is delayed as an outpatient
  Interventions: Procedure: Endoscopy

INTERVENTIONS:
Procedure: Endoscopy — Realization of an upper GI endoscopy

SUMMARY:
The purpose of this study is to validate the Glasgow-Blatchford score for the stratification of patients with upper gastro-intestinal hemorrhage. This score is easy to calculate. It is mainly based on the hemoglobin, blood pressure and blood urea. if the score is zero, the bleeding is very low risk and the gastrointestinal endoscopy may be delayed and performed as an outpatient.

ELIGIBILITY:
Inclusion Criteria:

* To be admitted in the university hospital for a gastrointestinal hemorrhage (vomiting of red or black blood or melena)

Exclusion Criteria:

* Age under 18
* Pregnancy
* Hemorrhage during hospitalisation
* red rectal bleeding
* No consent signed

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 208 (Actual)
Dates: Start 2009-10; Primary Completion 2010-06 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Comparison of length of stay between patients with score equal to zero and above zero | june 2010

SECONDARY OUTCOMES:
Determination of the proportion of low risk upper gastrointestinal bleeding | june 2010

CONTACTS AND LOCATIONS:
Overall Officials: Marc Girardin, MD, Principal Investigator — University Hospital, Geneva
Locations (1):
- Geneva University Hospital, Geneva, Switzerland

REFERENCES:
- [Background] Blatchford O, Murray WR, Blatchford M. A risk score to predict need for treatment for upper-gastrointestinal haemorrhage. Lancet. 2000 Oct 14;356(9238):1318-21. doi: 10.1016/S0140-6736(00)02816-6. PMID 11073021
- [Background] Stanley AJ, Ashley D, Dalton HR, Mowat C, Gaya DR, Thompson E, Warshow U, Groome M, Cahill A, Benson G, Blatchford O, Murray W. Outpatient management of patients with low-risk upper-gastrointestinal haemorrhage: multicentre validation and prospective evaluation. Lancet. 2009 Jan 3;373(9657):42-7. doi: 10.1016/S0140-6736(08)61769-9. Epub 2008 Dec 16. PMID 19091393